CLINICAL TRIAL: NCT00395772
Title: Once-daily Oral Direct Factor Xa Inhibitor BAY59-7939 in Patients With Acute Symptomatic Deep-vein Thrombosis The Einstein-DVT Dose-finding Study. A Phase II Evaluation.
Brief Title: Once-daily Oral Direct Factor Xa Inhibitor BAY59-7939 in Patients With Acute Symptomatic Deep-vein Thrombosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11528; EudraCT: 2004-002171-16
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Venous Thromboembolism
Keywords: Treatment of venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Arm 4 (Active Comparator)
  Interventions: Drug: (LMW) Heparin + Vitamin K Antagonist
- Arm 1 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)

INTERVENTIONS:
Drug: Xarelto (Rivaroxaban, BAY59-7939) — BAY59-7939 20 mg once daily (od) for 12 weeks
  Arms: Arm 1
Drug: Xarelto (Rivaroxaban, BAY59-7939) — BAY59-7939 30 mg od for 12 weeks
  Arms: Arm 2
Drug: Xarelto (Rivaroxaban, BAY59-7939) — BAY59-7939 40 mg od for 12 weeks
  Arms: Arm 3
Drug: (LMW) Heparin + Vitamin K Antagonist — Low Molecular Weight (LMW) Heparin + Vitamin K Antagonist (VKA) for 5 days, then VKA only for the rest of 12 weeks
  Arms: Arm 4

SUMMARY:
The purpose of this study is to determine the optimal dose of BAY 59-7939 and to compare the safety and effectiveness of this new drug with the standard way of treatment of deep vein thrombosis (heparin infusion plus one of the vitamin K antagonists), taking into account new events of thrombosis and pulmonary embolism and bleeding risk.

DETAILED DESCRIPTION:
Within the U.S., Johnson & Johnson is sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute symptomatic DVT, i.e. proximal or extensive calf-vein thrombosis involving at least the upper third part of the calf veins, without concomitant symptomatic PE
* Written informed consent

Exclusion Criteria:

* Legal lower age limitations (country specific)
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of DVT
* Other indication for VKA than PE/DVT
* More than 36 hours pre-randomization treatment with therapeutic dosages of (LMW) heparin or more than a single dose of VKA prior to randomization
* Participation in another pharmacotherapeutic study within the prior 30 days
* Creatinine clearance < 30 mL/min, impaired liver function (transaminases > 2 x ULN), or bacterial endocarditis
* Life expectancy < 3 months
* Active bleeding or high risk for bleeding contraindicating treatment with (LMW) heparin
* Uncontrolled hypertension: systolic blood pressure > 200 mmHg and diastolic blood pressure > 110 mmHg
* Pregnancy or childbearing potential without proper contraceptive measures
* Any other contraindication listed in the labeling of warfarin, acenocoumarol, phenprocoumon, fluindione, UFH, enoxaparin, or tinzaparin
* Systemic treatment with azole compounds or other strong CYP3A4 inhibitors (e.g. ketoconazole, fluconazol, itraconazole, HIV protease inhibitors) within 4 days prior to randomization and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2004-12; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the composite of symptomatic recurrent DVT or symptomatic fatal and non-fatal PE at 12 weeks and deterioration in thrombotic burden, as assessed by CUS and PLS, at baseline and at 12 weeks. | 12 weeks

SECONDARY OUTCOMES:
The principal safety outcome is all clinically relevant bleeding (i.e. major bleeding and clinically relevant non-major bleeding) within 12 weeks. | 12 weeks
The separate components of the primary efficacy outcome at 12 weeks. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (61):
- United States (4):
  - Albuquerque, New Mexico
  - Chapel Hill, North Carolina
  - Fredericksburg, Virginia
  - Seattle, Washington
- Australia (4):
  - Canberra, Australian Capital Territory
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Melbourne, Victoria
- Brazil (4):
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
- Canada (3):
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - London, Ontario
- Czechia (6):
  - Hradec Králové
  - Karlovy Vary
  - Ostrava
  - Pilsen
  - Prague
  - Ústí nad Labem
- Denmark (3):
  - Aarhus
  - Brædstrup
  - Frederiksberg
- France (6):
  - Brest
  - Grenoble
  - Montpellier
  - Paris
  - Saint-Etienne
  - Valenciennes
- Israel (9):
  - Afula
  - Ashkelon
  - Haifa
  - Holon
  - Kfar Saba
  - Petah Tikva
  - Safed
  - Tel Aviv
  - Tel Litwinsky
- Italy (5):
  - Milan
  - Padua
  - Pavia
  - Reggio Emilia
  - Venezia
- Netherlands (8):
  - Amersfoort
  - Amsterdam
  - Arnhem
  - Groningen
  - Hoofddorp
  - Maastricht
  - Sittard-geleen
  - Zwolle
- Poland (4):
  - Warsaw, Poland
  - Bydgoszcz
  - Warsaw
  - Wroclaw
- Johannesburg, Gauteng, South Africa
- Sweden (4):
  - Gothenburg
  - Jönköping
  - Stockholm
  - Västervik

REFERENCES:
- [Derived] Buller HR, Lensing AW, Prins MH, Agnelli G, Cohen A, Gallus AS, Misselwitz F, Raskob G, Schellong S, Segers A; Einstein-DVT Dose-Ranging Study investigators. A dose-ranging study evaluating once-daily oral administration of the factor Xa inhibitor rivaroxaban in the treatment of patients with acute symptomatic deep vein thrombosis: the Einstein-DVT Dose-Ranging Study. Blood. 2008 Sep 15;112(6):2242-7. doi: 10.1182/blood-2008-05-160143. Epub 2008 Jul 11. PMID 18621928
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/